CLINICAL TRIAL: NCT03210103
Title: A Randomized Trial of Treatment De-Escalation for HPV-Associated Oropharyngeal Squamous Cell Carcinoma: Radiotherapy vs. Trans-Oral Surgery (ORATOR II)
Brief Title: Primary Radiotherapy Versus Primary Surgery for HPV-Associated Oropharyngeal Cancer
Acronym: ORATOR2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ORATOR2
Record Dates: First submitted 2017-06-28; First posted 2017-07-06 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-12

CONDITIONS: Oropharyngeal Cancer
Keywords: Transoral Surgery; Head and Neck Cancer
MeSH Terms: conditions — Oropharyngeal Neoplasms; Head and Neck Neoplasms | interventions — Radiation; Drug Therapy; Neck Dissection

STUDY DESIGN:
Intervention Model Description: 2 Arm study randomized in a 1:1 ratio
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1, Radiation +/- Chemotherapy (Active Comparator): Standard Treatment (Radiation +/- Chemotherapy)
  Interventions: Radiation: Radiation
- Arm 2, TOS + Neck Dissection (Experimental): Transoral Surgery (TOS) + Neck Dissection (plus radiation, if required)
  Interventions: Procedure: Transoral Surgery (TOS) + Neck Dissection

INTERVENTIONS:
Radiation: Radiation — Standard of Care: Radiation +/- Chemotherapy
  Other Names: Chemotherapy, if required
  Arms: Arm 1, Radiation +/- Chemotherapy
Procedure: Transoral Surgery (TOS) + Neck Dissection — Transoral Surgery (TOS) + Neck Dissection (plus radiation, if required)
  Other Names: Radiation, if required
  Arms: Arm 2, TOS + Neck Dissection

SUMMARY:
The goal of this randomized treatment de-escalation study is to formally compare outcomes in HPV related oropharyngeal cancer tumors treated with a primary radiotherapy versus a primary surgical approach, to provide a high level of evidence to guide the selection of treatment options for a subsequent phase III trial

DETAILED DESCRIPTION:
The goal of this randomized treatment de-escalation study is to formally compare outcomes in HPV related oropharyngeal cancer tumors treated with a primary radiotherapy versus a primary surgical approach, to provide a high level of evidence to guide the selection of treatment options for a subsequent phase III trial

The study will compare overall survival rates relative to historical controls for de-intensified primary radiotherapy [60 GY +/- chemotherapy] versus transoral surgery (TOS) and neck dissection [+/- adjuvant 50Gy radiotherapy] in patients with early T-stage HPV-positive squamous cell carcinoma of the oropharynx and to compare quality of life (QOL) profiles.

The study will require a sample size of 140 patients randomized in a 1:1 ratio between the two arms. Arm 1 (radiotherapy +/1 chemotherapy) and Arm 2 (TOS)

Patients will be followed for a total of 5 years

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* willing to provide informed consent
* ECOG performance status 0-2
* Histologically confirmed squamous cell carcinoma
* P16 positive, or HPV positive
* Primary tumor site in the oropharynx (includes tonsil, soft palate, base of tongue, walls of oropharynx)
* Eligible for curative intent treatment, with likely negative resection margins at surgery. For patients where adequate transoral access is in question, they will first undergo an examination under anesthesia prior to randomization to ensure adequate exposure can be obtained.
* Smokers and non-smokers are included. Patients will be stratified by ,<10 pack years smoking history versus > or equal to 10 pack years.
* Tumor stage (AJCC 8th edition): T1 or T2
* Nodal stage (AJCC 8th edition): N0, N1, or N2
* For patients who may require chemotherapy (ie, patients with multiple lymph nodes positive or a single node more than 3 cm in size, in any plane, CBC/differential within 4 weeks prior to randomization with adequate bone marrow function, hepatic, and renal function defined as: Hemoglobin ≥ 80 g/L; Absolute neutrophil count ≥ 1.5 x 10 9/L, platelets ≥ 100 x 10 9/L, bilirubin ≤ 35 umol/L, AST or ALT ≤ 3 x the upper limit of normal; serum creatinine ≤ 130 umol/L or creatinine clearance ≥ 50 ml/min
* patients assessed at head and neck multidisciplinary clinic (with assessment by radiation oncologist and surgeon) and presented at multidisciplinary tumor board prior to randomization

Exclusion Criteria:

* unambiguous clinical or radiological evidence of extranodaal extension on pre-treatment imaging. This includes the presence of matted notes, defined as 3 or more nodes that are abutting with loss of intervening fat planes
* Serious medical comorbidities or other contraindications to radiotherapy, chemotherapy or surgery
* prior history of head and neck cancer within 5 years
* prior head and neck radiation at any time
* metastatic disease
* inability to attend full course of radiotherapy or follow up visits
* prior invasive malignant disease unless disease-free for at least 5 years or more, with the exception of non-melanoma skin cancer
* pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2018-01-26 (Actual); Primary Completion 2028-08-15 (Estimated); Study Completion 2028-08-15 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 2 years
  Time from randomization to death from any cause

SECONDARY OUTCOMES:
Quality of Life 1 year post treatment | 1 year post treatment
  Quality of life 1 year post treatment as assessed with the MD Anderson Dysphagia Inventory (MDADI)
Progression free survival comparison with historical controls | 5 years
  Defined as time from randomization to death from any cause
Quality of life | Baseline to 5 years follow up
  Quality of Life using the following questionnaire: MD Anderson Dysphagia Inventory (MDADI)
Quality of life | Baseline to 5 years follow up
  Quality of Life using the following questionnaire: EORTC QLQ C30
Quality of life | Baseline to 5 years follow up
  Quality of Life using the following questionnaire: H&N35 scale
Quality of life | Baseline to 5 years follow up
  Quality of Life using the following questionnaire: Voice Handicap Index (VHI-10)
Quality of life | Baseline to 5 years follow up
  Quality of Life using the following questionnaire: Neck Dissection Impairment Index (NDII)
Quality of life | Baseline to 5 years follow up
  Quality of Life using the following questionnaire: Patient Neurotoxicity Questionnaire (PNQ)
toxicity profile of both study arms using the National Cancer Institute Common Toxicity Criteria (NCI-CTC) Version 4 | Randomization until 5 years follow up
  To determine to toxicity profile of both study arms using the National Cancer Institute Common Toxicity Criteria (NCI-CTC) Version 4
Feeding tube rate at 1 year | baseline to 1 year post treatment
  Measure other functional measurements such as feeding tube rate at 1 year
CTCAE Dysphagia grade | baseline to 5 years post treatment
  Measure other functional measurements such as CTCAE Dysphagia grade
Speech intelligibility | baseline to 5 years post treatment
  Measure other functional measurements such as speech intelligibility
Normalcy of diet | baseline to 5 years post treatment
  Measure other functional measurements such as normalcy of diet
2 year progression-free survival comparison between Arm 1 and Arm 2 | 2 years
  Time from randomization to disease progress at any site or death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: David Palma, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (9):
- Australia (2):
  - Gold Coast University Hospital, Gold Coast, Queensland
  - Royal Adelaide Hospital, Adelaide
- Canada (7):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - BC Cancer, Vancouver, British Columbia
  - London Regional Cancer Program, London, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Sunnybrook Research Institute, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Palma DA, Prisman E, Berthelet E, Tran E, Hamilton S, Wu J, Eskander A, Higgins K, Karam I, Poon I, Husain Z, Enepekides D, Hier M, Richardson K, Mlynarek A, Johnson-Obaseki S, Gaudet M, Bayley A, Dowthwaite S, Jackson JE, Dzienis M, O'Neil J, Chandarana S, Banerjee R, Hart R, Chung J, Tenenholtz T, Le H, Yoo J, Mendez A, Winquist E, Kuruvilla S, Stewart P, Warner A, Mitchell S, Chen J, Parker C, Kwan K, Theurer J, Bahig H, Christopoulos A, Mendez LC, Sathya J, Hammond JA, Read N, Venkatesan V, Fung K, Nichols AC. Radiation vs. trans-oral surgery for treatment de-escalation in HPV-related oropharyngeal cancers: Primary analysis of the ORATOR2 randomized trial. Eur J Cancer. 2025 May 2;220:115343. doi: 10.1016/j.ejca.2025.115343. Epub 2025 Mar 10. PMID 40121836
- [Derived] Palma DA, Prisman E, Berthelet E, Tran E, Hamilton S, Wu J, Eskander A, Higgins K, Karam I, Poon I, Husain Z, Enepekides D, Hier M, Sultanem K, Richardson K, Mlynarek A, Johnson-Obaseki S, Odell M, Bayley A, Dowthwaite S, Jackson JE, Dzienis M, O'Neil J, Chandarana S, Banerjee R, Hart R, Chung J, Tenenholtz T, Krishnan S, Le H, Yoo J, Mendez A, Winquist E, Kuruvilla S, Stewart P, Warner A, Mitchell S, Chen J, Parker C, Wehrli B, Kwan K, Theurer J, Sathya J, Hammond JA, Read N, Venkatesan V, MacNeil SD, Fung K, Nichols AC. Assessment of Toxic Effects and Survival in Treatment Deescalation With Radiotherapy vs Transoral Surgery for HPV-Associated Oropharyngeal Squamous Cell Carcinoma: The ORATOR2 Phase 2 Randomized Clinical Trial. JAMA Oncol. 2022 Jun 1;8(6):1-7. doi: 10.1001/jamaoncol.2022.0615. PMID 35482348
- [Derived] Nichols AC, Lang P, Prisman E, Berthelet E, Tran E, Hamilton S, Wu J, Fung K, de Almeida JR, Bayley A, Goldstein DP, Eskander A, Husain Z, Bahig H, Christopoulous A, Hier M, Sultanem K, Richardson K, Mlynarek A, Krishnan S, Le H, Yoo J, MacNeil SD, Mendez A, Winquist E, Read N, Venkatesan V, Kuruvilla S, Warner A, Mitchell S, Corsten M, Rajaraman M, Johnson-Obaseki S, Eapen L, Odell M, Chandarana S, Banerjee R, Dort J, Matthews TW, Hart R, Kerr P, Dowthwaite S, Gupta M, Zhang H, Wright J, Parker C, Wehrli B, Kwan K, Theurer J, Palma DA. Treatment de-escalation for HPV-associated oropharyngeal squamous cell carcinoma with radiotherapy vs. trans-oral surgery (ORATOR2): study protocol for a randomized phase II trial. BMC Cancer. 2020 Feb 14;20(1):125. doi: 10.1186/s12885-020-6607-z. PMID 32059705